CLINICAL TRIAL: NCT00791453
Title: Clarksdale Diabetes and Metabolism Clinic Consumer Health Education Center Study
Brief Title: Clarksdale Diabetes and Metabolism Clinic CHEC Study
Acronym: CHEC
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Jacinda Roach/Assistant Professor, Deptartment of Medicine,, The University of Mississippi Medical
Other Study IDs: 2008-0001; NO1-LM-6-3502
Record Dates: First submitted 2008-01-28; First posted 2008-11-14 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes
Keywords: Diabetic patients at the Clarksdale Diabetes; and Metabolism Clinic and must be between the; ages of 18 and 64 years of age.
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No biospecimens are retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Established patients at the Clarksdale Diabetes and Metabolism Center
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Patients will receive literacy appropriate health information.

SUMMARY:
This study will involve established clinic patients. The Rapid Estimate of Adult Literacy in Medicine will be administered during patients' regular clinic visits. Patients will then be referred to the Consumer Health Education Center (CHEC)by healthcare providers who will fill out a referral form. The form will be given the the CHEC health educator who will assist patients in finding literacy-appropriate health information. BMI and Hgb A1c values will be compared after 3 months and 6 months to baseline values. It is hypothesized that objective assessment of patient use of literacy-appropriate, health information from the Clarksdale Diabetes and Metabolism Clinic CHEC will improve Hgb A1c and BMI values among patients.

ELIGIBILITY:
Inclusion Criteria:

* Established patients of the Clarksdale Diabetes and Metabolism Clinic between the ages of 18 and 64.

Exclusion Criteria:

* Individuals who are not established patients of the clinic and are not between the ages of 18 and 64.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Established patients at a diabetes clinic.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Hgb A1C and BMI measurements will improve | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacinda B. Roach, PhD, Principal Investigator — The University of Mississippi Medical Center
Locations (1):
- The University of Mississippi Medical Center, Jackson, Mississippi, United States